#### **QUESTIONNAIRE**

**Date:** 4<sup>th</sup> September 2021

**Version:** Version 3

Title: Patterns and risk factors for suicide ideation among in-school adolescents in Nigeria

and a comprehensive suicide-behavior prevention intervention pilot study

Researcher: ABIODUN, Olumide Adetokunbo

**Institution:** ICT University Cameroon/University of Turku, Finland

Purpose: In partial fulfillment of the requirements for the award of Ph.D. Epidemiology

#### PARTICIPANTS' CONSENT FORM

| Dear Ms./Mr |
|-------------|

I invite you to participate in this research. I am Dr. Olumide ABIODUN a Ph.D. Candidate of the ICT university, Cameroon and the Injury Epidemiology and Prevention (IEP) Research Group, Turku Brain Injury Centre University of Turku, Turku, Finland. I am conducting a research for my doctoral thesis.

Please read/listen to the reading of this document carefully. It provides important information to help you decide whether or not to participate in this research. Local staff members of research are also available to give you more details. You should feel free to ask any questions or discuss any concerns. Your participation is completely voluntary. Even after deciding to participate, you may withdraw at any time. There will be negative consequences if you choose not to participate or withdraw from the study at any time.

#### General information about the Study

#### Why are we doing this study?

In order to best understand and mitigate the results of behaviors related to suicide, especially suicide thought among adolescents, there is a need to assess the burden and determinants of suicidal ideation. This study will help characterize the experience of suicide ideation, its risk and protective factors.

# Who will participate in this research?

We are recruiting 1440 young people between the ages of 10 and 19 years who are currently enrolled in secondary schools. They will be interviewed to assess suicide thoughts and the factors that are related to it.

# What does my participation involve?

The study will take place in ten secondary schools spread around Ogun State, Nigeria over six months. Each consenting participant is required to answer some questions. The interview should last between 40 and 45 minutes. A study staff will guide each participant through the interview process. They will advise and address your concerns. Your names or personal identification details will not be requested. Data collection will be done in a private room to make you comfortable and prevent others listening to your answers.

# What will you do with my responses?

Your responses will be used for research purposes and to advise policy Your data and sample may be shared with other researchers for further study purpose only. Your unique identifier will not be requested or shared for any purpose whatsoever. All such all information got from you will remain confidential.

# Where will my data be stored?

Your data will be kept securely by the investigator. Those to whom the data will be shared will be required to sign an agreement for the ethical use of data.

#### What if I decide not to participate in the study?

If you do not wish to participate in this study, no one will treat you differently. Declining will not cause you to lose any benefits you have been receiving in school. Your teachers will not change towards you. You can withdraw from the study at any time without giving any explanation. Withdrawing will not cause any problems for you. If you leave the study, you can request that your data not be used in future analyses. At your request, we will destroy any data still controlled by the investigator but may not be able to destroy data given to other researchers.

# Is there any risk or inconvenience for those who participate in this study?

The interview will take some time and may involve answering some very personal questions.

# Will it cost me anything?

There is no financial cost to you for participating in this study.

# What benefit do I get?

The results of the investigation will be used make advocacy and advise policy towards improving the mental health of adolescents. Participants will be free to ask questions about the subjects and should expect the questions to be answered.

# Will I receive compensation for my participation in this study? No.

# To whom should I direct any questions?

If you have additional questions or wish to withdraw your participation in the future, please the investigators, Dr. Olumide ABIODUN on +234 703 856 9725

# **Declaration of consent:**

**Ethics Committee approval date:** 

**Duration of Ethics Committee approval:** 

I understand that my signature verifies that I have read this information. I agree to participate in the study. I acknowledge receiving a signed copy of this document.

| Participant Signature: | |
|---|---|
| Name (Print): Declaration of Assent: | Date: |
| I hereby give assent for my child/ward to participate in Parent/Guardian Signature: | |
| Name (Print): | Date: |
| Statement by the researcher/person taking consent I have accurately read out the information sheet to the potential participant, and to the best of my ability made sure that the participant understands what will be done I confirm that the participant was given an opportunity to ask questions about the study, and all the questions asked by the participant have been answered correctly and to the best of my ability. I confirm that the individual has not been coerced into giving consent, and the consent has been given freely and voluntarily. A copy of this informed consent form has been provided to the participant. Name of person taking the consent: Signature of person taking the consent: | |
| Date: | |
| Ethics Committee assigned approval number: | BUHREC001/21 |

1st February, 2021

Not applicable